CLINICAL TRIAL: NCT06842589
Title: Study of Therapeutic Efficacy of Anti-CD19 Chimeric Antigen Receptor T Lymphocytes (CAR-T) Cells in Patients With Multi-drug Resistant SRNS
Brief Title: Study of Therapeutic Efficacy of Anti-CD19 CAR-T Cell Therapy in Patients With MDR-SRNS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SC-0001-P-01
Record Dates: First submitted 2025-01-22; First posted 2025-02-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: Multi-Drug Resistant Nephrotic Syndrome; CAR-T Cell Therapy
Keywords: car-t; Multi-Drug Resistant Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T treatment group (Experimental): This study employs a '3+3' design with three dosage groups (0.3×10^5/kg, 1×10^5/kg, and 3×10^5/kg). Each dosage group will enroll 3 to 6 patients, starting from the lowest dosage and escalating to explore a safe and effective dose. Once a dosage group completes enrollment without observing any serious unexpected adverse reactions, and based on the efficacy and cell kinetics data, the investigator and the technical team together may consider escalating to the next dosage group to explore the optimal effective dose. The trial is expected to enroll a total of 9 to 18 patients
  Interventions: Biological: anti-CD19 CAR-T cells

INTERVENTIONS:
Biological: anti-CD19 CAR-T cells — Three dose groups (0.3×105/kg, 1×105/kg, 3×105/kg) were set up, starting from the low dose group climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of anti-CD19 CAR-T cells in the treatment of patients with Multi-drug resistant SRNS

DETAILED DESCRIPTION:
At present, there is no effective treatment for Multi-drug resistant steroid resistant nephrotic syndrome (MDR-SRNS), which has a high risk of progression to kidney failure, and about 55% of patients will have disease recurrence after receiving kidney transplantation, which is in urgent need of new treatment methods.

CAR-T therapy is an adoptive cell therapy that uses genetic modification technology to reprogram T cells and eliminate target cells expressing disease-related antigens through antigen-specific recognition.Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases. Although no clinical data related to CAR-T treatment of nephrotic syndrome has been disclosed, CAR-T is effective for systemic lupus erythematosus and systemic sclerosis.Many kinds of autoimmune diseases such as chemical syndrome and idiopathic inflammatory dermatomyositis have good therapeutic effect. These results suggest that the therapeutic effect of CAR T cells may not be limited to systemic lupus erythematosus, but may also play a role in several different B-cell-mediated and autoantibody-driven human autoimmune diseases, which is expected to bring breakthroughs in the treatment of MDR-SRNS.The purpose of this study is to assess the safety and efficacy of the anti-CD19 CAR-T cells in the treatment of patients with MDR-SRNS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥2 years old, gender unlimited;
* 2.Diagnosed with SRNS according to the 2021 Kidney Disease: Improving Global Outcomes （KDIGO） Guidelines and have not achieved a complete response after 12 months of treatment with two standard doses of hormone replacement drugs with different mechanisms of action or relapse of disease activity after remission (at least one of the two drugs is a calcineurin inhibitor such as cyclosporine or tacrolimus; Other hormone replacement drugs include Mycophenolate Mofetil, cyclophosphamide, Taitacept or rituximab); Or if no remission has been achieved after 3 to 6 months of adequate treatment with one calcineurin inhibitor, if the researcher judges that the benefits outweigh the risks and the patient or guardian has fully informed consent, the patient can be considered for inclusion.Patients with other diseases, such as systemic lupus erythematosus, requiring long-term systemic treatment with glucocorticoids or immunosuppressants, may be considered for inclusion after the investigator determines that the benefits outweigh the risks and the patient or guardian has fully informed consent;
* 3. Renal biopsy was performed and the pathological type was determined to be minimal lesion nephropathy(MCD) or focal segmental glomerulosclerosis (FSGS);
* 4. The functions of important organs are basically normal: Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% with no obvious abnormality in electrocardiogram; Renal function: eGFR≥30ML/min/1.73m2# Liver function: Asparagus cochinchinensis transaseminase (AST) and Alanine Aminotransferase (ALT)≤3.0 upper limit of normal, Total Bilirubin (TBIL) in serum ≤2.0×upper limit of normal; Lung function: No serious lung lesions, SpO2≥92%;
* 5. Met the standards of leukapheresis or intravenous blood collection, No contraindication for cell collection;
* 6. Negative pregnancy test for female Subjects of childbearing age, agree to take effective contraceptive measures the first year after CAR-T infusion;
* 7. Participants or their guardians agrees to participate in the clinical trial and sign the informed consent form which indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

* 1. Received CAR T cell therapy or other gene-modified cell therapy previously;
* 2. Patients had a cerebrovascular accident or seizure, or other active central nervous system disease within 6 months;
* 3. Genetic tests have confirmed hereditary kidney disease;
* 4. Renal biopsy has been confirmed as immunoglobulin A nephropathy, idiopathic membranous nephropathy or membranoproliferative glomerulonephritis;
* 5. Renal replacement therapy has been or is being performed within 3 months prior to transfusion. (if acute kidney injury factors were considered, patients with chronic kidney disease were excluded, and the benefits outweighed the risks as determined by the investigator and with the full and informed consent of the patient or guardian could be considered for inclusion);
* 6. Renal replacement therapy has been or is being performed within 3 months prior to transfusion;
* 7. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs;
* 8. Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months prior to screening; Acute graft-versus-host disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening;
* 9. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
* 10. Macrophage activation syndrome occurred within 1 month prior to screening;
* 11. Received live vaccine within 4 weeks before screening;
* 12. Patients with malignant diseases such as tumors before screening, or with other serious life-threatening diseases;
* 13. Tested positive in Blood pregnancy test;
* 14. Patients who participated in other clinical study within 1 months prior to enrollment;
* 15. Any other conditions that the investigators deem it unsuitable for the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-14 (Estimated); Primary Completion 2027-02-14 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR-T cell therapy in patients with MDR SRNS | 3 months
  Incidence and severity of Adverse Events (AEs) and Serious Adverse Event（SAEs）,including changes in laboratory values,Electrocardiograph(ECG) and vital signs assessed by CommonTerminology Criteria for Adverse Events (CTCAE) v5.0.
The efficiency of CAR-T cell therapy in patients with MDR SRNS | 3 months
  Complete response and partial response rate (complete response defined as Urinary protein/creatinine ratio (uPCR) ≤200 mg/g for 3 consecutive days, partial response is defined as a 50% or more reduction in proteinuria from baseline and 200mg/g < uPCR <2000mg/g)

SECONDARY OUTCOMES:
Effectiveness of other visit points | 24 months
  Rate of complete or partial response at other visit points after cell infusion (1 month, 2 months, 6 months, 9 months, 12 months, 18 months, 24 months)
Pharmacokinetic Outcome Cmax | 3 months
  The highest concentration (Cmax) of targeted CD19 CAR-T cells expanded in peripheral blood after infusion
Pharmacokinetic Outcome Tmax | 3 months
  The time to reach the maximum concentration (Tmax)
Pharmacokinetic Outcome AUC | 3 months
  The area under the curve (AUC) at 28 days and 90 days post-infusion (AUC28d/90d)
Pharmacodynamics Outcome | 3 months
  The degree of B cell clearance at various time points, and the concentration levels of CAR-T related serum cytokines such as IL-6, CRP, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No